CLINICAL TRIAL: NCT02014831
Title: A Randomized Phase II Study to Evaluate the Efficacy and Safety of Cetuximab in Metastatic Penile Carcinoma
Brief Title: Efficacy and Safety of Cetuximab in Metastatic Penile Carcinoma (PENILANE)
Acronym: PENILANE
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Industry decline to supply study drug
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PENILANE
Record Dates: First submitted 2013-12-05; First posted 2013-12-18 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2016-02

CONDITIONS: Squamous Cell Carcinoma of the Penis
Keywords: Squamous Cell Carcinoma of the penis; Stage N3; Metastasis; TIP; Cetuximab; Objective Response Rate; Safety profile; Overall Survival; Progression Free Survival; Quality of Life
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TIP (Active Comparator): "Reference" arm; Patients will be treated with 6 cycles of Paclitaxel + Ifosfamide + Cisplatin (TIP treatment)
  Interventions: Drug: TIP
- Cetuximab + TIP (Experimental): "Experimental" arm: Patients will be treated with 6 cycles of Paclitaxel + Ifosfamide + Cisplatin (TIP treatment) and weekly infusion of Cetuximab.
  Interventions: Drug: Cetuximab; Drug: TIP

INTERVENTIONS:
Drug: Cetuximab — Cetuximab treatment will be administered on specific days within a 21-days-cycle and for a maximum of 6 cycles as follow :
  CETUXIMAB I.V infusion of 400 mg/m2 on cycle 1 Day 0 for 2 hours, then 250 mg/m2 for subsequent infusions for 1 hour on Day 8, Day 15 and next cycles Day1, Day8, Day15.
  In case of documented toxicities, 2 drugs doses reductions are allowed according specific algorithms indicated in protocol
  Arms: Cetuximab + TIP
Drug: TIP — The TIP combination of treatments will be administered on specific days within a 21-days-cycle and for a maximum of 6 cycles as follow :
  PACLITAXEL I.V infusion of 175 mg/m2, for 3 hours, on Day 1 of the cycle.
  IFOSFAMIDE I.V infusion of 1200 mg/m2, for 2 hours, on Day 1, Day 2, Day 3 of the cycle.
  CISPLATINE I.V infusion of 25 mg/m2, for 1 hour, on Day 1, Day 2, Day 3.
  In case of documented toxicities, 2 drugs doses reductions are allowed according specific algorithms indicated in protocol

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Cetuximab in metastatic penile carcinoma

DETAILED DESCRIPTION:
Penile carcinoma is a rare cancer type, particularly in our industrialized countries. Incidence is not well established but is estimated around 26000 annual new cases all around the world [1]. We don't have accurate estimation for France but regarding data from the literature, incidence rates in developed countries vary from 0.7 to 1.0/100000 men [2]. The mean age at diagnosis is about 60 years [3].

Different causes have been identified like history of Human PapillomaVirus (essentially HPV16), phymosis, absence of circumcision, tobacco use, and history of condyloma [1]. In addition, a lot of molecular genetic alterations are also responsible for penile cancer occurrence and development [4].

Histologically, most of these tumors are epidermoid cancers. Tumor spreads into inguinal lymphnodes, then into pelvic lymphnodes. Then retroperitoneal lymphnodes are involves before metastatic dissemination, often in lungs, liver and bones.

According to the French urology recommendations, treatment of localized penis cancer should be conservative, as far as possible [5]; Even if local recurrences rate varies from 15% to 30% of patients, no reduction of overall survival is observed in these patients [7].

The investigations regarding involvement of inguinal lymphnodes and distant organs are a key-point. Among the 10% of patients with loco regional recurrence [6], lymphadenectomy should be preferred to chemotherapy which should be recommended for metastatic patients or unresectable patients with regional lymphnodes involvement [5].

Numbers of treatments (monotherapy or associations) have been tested in penis cancer but the rarity of these tumors is a major obstacle to clinical research, due to small samples of patients. The best results seem to be obtained with platinum-based treatments (ORR up to 32.5% with a combination of cisplatin, methotrexate and bleomycine) [8] [9], but even if response rates are very promising, overall survival is still very short (median OS = 28 weeks) and treatment-related toxicities can be very important, even lethal [9].

The histological type of squamous cells carcinoma, which is the large majority of penile cancer, led Pagliaro et al. [10] to explore a combination of Paclitaxel, Ifosfamide and Cisplatin (TIP) as neoadjuvant treatment of locally advanced penile tumors. This association of chemotherapy agents had previously proven its efficacy in squamous cell carcinoma of the head and neck. Even if this study included a small number of patients (N=30) with penile carcinoma, it showed very promising results on primary objective (objective response rate = 50% with 10% of complete responses).

Despite these results and all previous researches, no chemotherapy agent has been submitted to health authority's approval in France. It results that there is no market approval for treatment of metastatic penile carcinoma.

However, based on the results of Pagliaro et al., the TIP is now considered by the French physicians as the recommended standard of care for patients with metastatic penile carcinoma [5].

From a biological point of view, Epidermal Growth Factor Receptor (EGFR) and K-ras status have been widely explored in the past few years in penile carcinoma.

EGFR seem to present high expression levels in such tumors, whatever the stage of disease. Among 17 patients studied by Lavens et al., expression of EGFR was 3+ (which is the highest grade of expression) in 14 cases and 2+ in 3 cases [11].

Andersson et al. analyzed 28 penis tumors and found a somatic mutation in 39% (n=11). Mutations have been detected in the following genes: PIK3CA (29%), HRAS (7%) and K-ras (3%) [12].

Dorff et al. studied EGFR expression and K-ras status in 28 other penile carcinomas. They noted an over expression of EGFR in all the samples but didn't find any K-ras mutation [13] while Valverde et al. found 22% of K-ras muted carcinomas (N=28) [14].

When present, K-ras mutations have been identified on exon 2 (codons 12 and 13) but rarely on exon 3 (codon 61). Mutational status can be easily explored by Polymerase Chain Reaction amplification.

EGFR expression seems to be correlated with differentiation grade while K-ras mutation seems to be correlated to the stage of disease [13] [14].

Cetuximab is a human/mouse chimeric monoclonal antibody. It has a specific and competitive binding to the extracellular domain of EGFR, leading to inactivation of self-phosphorylation of the receptor and inhibition of all the following intracellular signal chains. This has an antiproliferative effect on cancer cells, inhibits angiogenesis, reduces cells mobility and restores apoptosis.

Cetuximab has been widely studied in cancers with overexpression of Epidermal Growth Factor Receptors (EGFR), in particular in squamous cancers of head and neck [15], colorectal [16] and lung cancers [17].

Phases I studies showed that a dose in the range of 200mg/m² to 400mg/m² led to a good EGF receptor saturation [18]. Association of Cetuximab and radiation therapy showed an improvement on overall survival in patients with locally advanced head and neck cancers (median overall survival = 49 months versus 29 months in the radiotherapy-alone group) [19].

Cetuximab has also been associated to platinum-based chemotherapies (Cisplatin or Carboplatin) and 5-Fluorouracile in patients with head and neck cancer. Median overall survival was significantly better on the group of patients with Cetuximab (10.1 months vs 7.4 months; p=0.04). However, 82% of patients with Cetuximab experienced Commom Terminology Criteria for Adverse Event (CTCAE) grade 3/4 toxicities versus 76% in the other group [20].

Adverse events commonly noted with Cetuximab are cutaneous events, hypomagnesaemia, infection and grade 3/4 anorexia.

Cetuximab has also been studied as monotherapy in head and neck patients with responses rate of 13% and disease control rate of 46%. Cutaneous events were still the main toxicities [21].

One preliminary experience has been conducted in a patient with penile carcinoma, treated with an association of a taxane (Docetaxel) and Cetuximab. This treatment led to imaging and clinical signs of efficacy (decrease of 18F-2-fluoro-2-deoxy-D-glucose fluorodeoxyglucose (18-FDG) uptake, necrosis of metastatic mass, improvement of pain and performance status). The tolerance profile has been characterized by neutropenia and mild skin toxicity [22].

Another key-point is that the efficacy of Cetuximab is closely related to the presence of mutation on the gene coding for K-ras. Van Cutsem et al. showed that patients with wild-type K-ras colorectal cancers are much better responders to Cetuximab than patients with mutation [23].

K-ras mutation leads to a constitutive activation of the Ras pathway independently and can bypass the EGFR-driven signaling cascade and impair the clinical efficacy of EGFR.

K-ras status should always be determined before Cetuximab initiation and it would be interesting to know EGFR expression rates in order to correlate with responses to Cetuximab.

Finally, immunogenicity is a class effect of monoclonal chimeric antibodies; the incidence of Human Anti-Chimeric Antibodies (HACA) formation has been observed around 3.7% of patients treated with cetuximab. However, no apparent effect on the safety or antitumor activity of cetuximab has been observed in these patients [Summary of Product Characteristics of Cetuximab].

Given the fact that,

* the association of Paclitaxel, Ifosfamide and Cisplatin is efficient for the treatment of metastatic penile carcinoma and considered as the new "standard" of care in France,
* squamous cell carcinoma of the penis expresses EGF receptor,
* cetuximab has anti-tumor properties in EGF mediated cancers,
* response rates to cetuximab is much better in patient with wild-type K-ras,

We postulate that:

- the combination of Paclitaxel, Ifosfamide, Cisplatin with Cetuximab, will enable to provide a better Objective Response Rate (ORR) than the same combination used without Cetuximab.

As promising results obtained by Pagliaro are not resulting from a comparative phase III with a reference treatment, it cannot be considered as a validated new standard of care.

The proposed Phase 2 study will explore the optimal way to treat patients with metastatic penile carcinoma between two experimental schemes using a Simon's selection "pick the winner" randomized design.

ELIGIBILITY:
INCLUSION CRITERIA :

* Male older than 18 years-old,
* Squamous cell carcinoma of the penis of clinical stages N3 and/or M1,
* Central Histological confirmation of diagnosis of wild-type K-ras penis cancer (histological documentation of the mutational status prior to each patient's registration).

Nota Bene: an archival tumor sample must be available.

* At least one measurable lesion according to the RECIST version 1.1. In case of relapsing patient, documented progression as per RECIST version 1.1,
* Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 2,
* Life expectancy ≥ 6 months,
* Adequate organs functions defined as the following (transfusion is not allowed within 7 days prior to lab test performed to assess the eligibility):

  * Hemoglobin ≥ 9 mg/dL,
  * Absolute Neutrophils Count ≥ 1,5 Gi/l,
  * Platelets ≥ 100 Gi/l,
  * Creatinine ≤ 1,5 x Upper Limit of Normal (ULN) and Creatinine clearance ≥ 60 ml/min (calculated with Cockcroft formula or Modification of Diet in Renal Disease (MDRD) formula for patients older than 65 years old)
  * Aspartate aminotransferase (ASAT) and Alanine aminotransferase (ALAT) ≤ 2,5 x ULN (≤ 5 x ULN in presence of liver metastasis)
  * Total bilirubin ≤ 1,5 x ULN,
* Willingness to use effective contraceptive method during the whole treatment period and up to 4 months after the last study drug administration,
* Affiliated to the French social security system,
* Subjects must provide written informed consent prior to perform any study-specific procedures or assessments and must be willing to comply with treatment and follow up.

EXCLUSION CRITERIA :

* Symptomatic metastases of Central nervous system (CNS) requiring or having required steroids or enzyme-inducing anticonvulsants within 4 weeks before inclusion,
* Previous treatment with paclitaxel, or ifosfamide, or cetuximab, or any monoclonal antibody, and or any drug targeting EGF Receptor,
* Local and/or resectable disease,
* Prior history of other malignancies other than penis cancer (except for basal cell or squamous cell carcinoma of the skin and superficial bladder carcinoma) unless the subject has been free of the disease for at least 3 years,
* No resolution of specific toxicities related to any prior anti-cancer therapy to Grade ≤1 according to the CTCAE v.4.0 (except lymphopenia and alopecia),
* Active peripheral or motor neuropathy of any CTCAE grade and due to any cause,
* Known hypersensitivity or allergy or contraindication to at least one of the study drugs
* In case of previous chemotherapy, wash out period of less than 5 half-lives of treatment before study entry,
* Clinically significant cardiovascular disease including:

  * Myocardial infarction within 3 months,
  * Congestive heart failure of the New York Heart Association (NYHA) class 3 or 4, or patients with history of congestive heart failure NYHA class 3 or 4 in the past, unless a screening Left Ventricular Ejection Fraction (LVEF) assessment ≥ 45%,
  * Prolonged QT interval defined as screening corrected QT interval (QTc) > 470 ms (Fridericia correction formula),
  * History of clinically significant ventricular arrhythmia (e.g., ventricular tachycardia, ventricular fibrillation, ...),
  * History of Mobitz II 2nd degree or 3rd degree heart block without a permanent pacemaker in place,
  * Hypotension (systolic BP < 86 mmHg) or bradycardia with a heart rate < 50 bpm,
  * Uncontrolled hypertension as indicated by a resting systolic BP > 170 mmHg or diastolic BP > 105 mmHg despite an optimal treatment,
* Major surgery or radiation therapy within 4 weeks prior first study drug administration or already planned during the study,
* Any pulmonary, thyroid, renal, hepatic severe/uncontrolled concurrent medical disease that in the opinion of the investigator could cause unacceptable safety risks or compromise compliance with the protocol,
* Active uncontrolled viral, fungal or bacterial infection,
* Patient who cannot abstain from vaccine against yellow fever, prophylactic use of phenytoin or derivate, or any drug which can strongly interfere with the sub-units 2C8 and/or 3A4 of the cytochrome P450 (Cf. appendix 5) Nota Bene: in case of poor interference with these sub-units, treatments with a narrow therapeutic index should be avoided.
* Active drug or alcohol use or dependence that, in the opinion of the investigator, would interfere with adherence to study requirements (participants must agree to refrain from substance abuse use during the entire course of the study),
* Concomitant participation to another clinical trial with active agent during the study (concomitant non interventional study will be allowed).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-02; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Evaluation of the antitumor activity of Cetuximab treatment in terms of Objective Response Rate (ORR) at the end of treatment | 4 weeks after the day 1 of the last cycle administered (i.e between 4 weeks to 20 weeks after randomization, according to the amount of administered cycles)
  Patients will be treated by TIP +/- Cetuximab for 1 cycle of 21 days. Subsequent treatment cycles will be performed only if patients meet correct biological analyses as defined by protocol, with a maximum of 5 more cycles of 21 days. Thus, the treatment duration will vary between patients from 3 weeks to 18 weeks. The treatment efficacy will be evaluated 28 days after the day 1 of the last cycle administered. Thus ORR will be evaluated between 4 weeks to 20 weeks after randomization, according to the amount of administered cycles.
  ORR is defined as the proportion of patients with best response consisting in a Complete Response (CR) or a Partial Response (PR) from the date of randomization to the date of the end of treatment visit (i.e 6 cycles of treatment as maximum) evaluated according to the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1

SECONDARY OUTCOMES:
Evaluation of the Safety Profile of Cetuximab treatment | From patient randomization up to the end of study i.e 28 months maximum after first patient inclusion
  Safety profile is assessed throughout the study by incidence and intensity of Adverse Events displayed by patients using the CTCAE version 4.0
Evaluation of the antitumor activity of Cetuximab treatment in terms of Overall Survival (OS) at the end of the study | From patient randomization up to the end of study i.e 28 months maximum after first patient inclusion
  OS is defined as the time from the date of randomization to the date of death due to any cause. If a patient is not known to have died at the time of the analysis, OS will be censored at the date of last contact.
Evaluation of the antitumor activity of Cetuximab treatment in terms of Progression-Free Survival (PFS) at the end of the study | From patient randomization up to the end of study i.e 28 months maximum after first patient inclusion
  PFS is defined as the time from the date of randomization to the date of event defined as the first documented progression or death due to any cause. If a patient has not had an event at the time of the analysis, PFS will be censored at the date of last adequate tumor assessment.
Evaluation of Quality of Life during the Cetuximab treatment | From patient randomization up to the end of treatment (i.e between 4 weeks to 20 weeks after randomization, according to the amount of administered cycles)
  Quality of life is assessed using the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) C30. It will be evaluated at Screening, at the beginning of cycle 4, and at the end of treatment i.e after 6 cycles maximum

CONTACTS AND LOCATIONS:
Overall Officials: Helen BOYLE, Doctor, Principal Investigator — Centre Leon Berard
Locations (7):
- France (7):
  - CHRU Strasbourg, Strasbourg, Bas Rhin
  - Institut Paoli Calmettes, Marseille, Bouches du Rhône
  - Institut Bergonié, Bordeaux, Gironde
  - Institut Claudius Regaud, Toulouse, Haute Garonne
  - Centre Léon Bérard, Lyon, Rhône
  - Institut Curie, Paris, Île-de-France Region
  - APHP Hôpital Saint Louis, Paris, Île-de-France Region

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bleeker MC, Heideman DA, Snijders PJ, Horenblas S, Dillner J, Meijer CJ. Penile cancer: epidemiology, pathogenesis and prevention. World J Urol. 2009 Apr;27(2):141-50. doi: 10.1007/s00345-008-0302-z. Epub 2008 Jul 8. PMID 18607597
- [Background] Barnholtz-Sloan JS, Maldonado JL, Pow-sang J, Giuliano AR. Incidence trends in primary malignant penile cancer. Urol Oncol. 2007 Sep-Oct;25(5):361-7. doi: 10.1016/j.urolonc.2006.08.029. PMID 17826651
- [Background] Curado M.P., Edwards B., Shin H.R. et al. Cancer Incidence in Five continents. Sci Publ. 2007. 160:570-573.
- [Background] Calmon MF, Tasso Mota M, Vassallo J, Rahal P. Penile carcinoma: risk factors and molecular alterations. ScientificWorldJournal. 2011 Feb 3;11:269-82. doi: 10.1100/tsw.2011.24. PMID 21298218
- [Background] Rigaud J., Avancès C., Camparo P. et al. Recommendations en onco-urologie 2010: Tumeurs malignes du penis. Progrès en oncologie. 2010. Suppl.4:279-289.
- [Background] Philippou P, Shabbir M, Malone P, Nigam R, Muneer A, Ralph DJ, Minhas S. Conservative surgery for squamous cell carcinoma of the penis: resection margins and long-term oncological control. J Urol. 2012 Sep;188(3):803-8. doi: 10.1016/j.juro.2012.05.012. Epub 2012 Jul 19. PMID 22818137
- [Background] Smith Y, Hadway P, Biedrzycki O, Perry MJ, Corbishley C, Watkin NA. Reconstructive surgery for invasive squamous carcinoma of the glans penis. Eur Urol. 2007 Oct;52(4):1179-85. doi: 10.1016/j.eururo.2007.02.038. Epub 2007 Feb 20. PMID 17349734
- [Background] Di Lorenzo G, Buonerba C, Federico P, Perdona S, Aieta M, Rescigno P, D'Aniello C, Puglia L, Petremolo A, Ferro M, Marinelli A, Palmieri G, Sonpavde G, Mirone V, De Placido S. Cisplatin and 5-fluorouracil in inoperable, stage IV squamous cell carcinoma of the penis. BJU Int. 2012 Dec;110(11 Pt B):E661-6. doi: 10.1111/j.1464-410X.2012.11453.x. Epub 2012 Sep 10. PMID 22958571
- [Background] Haas GP, Blumenstein BA, Gagliano RG, Russell CA, Rivkin SE, Culkin DJ, Wolf M, Crawford ED. Cisplatin, methotrexate and bleomycin for the treatment of carcinoma of the penis: a Southwest Oncology Group study. J Urol. 1999 Jun;161(6):1823-5. PMID 10332445
- [Background] Pagliaro LC, Williams DL, Daliani D, Williams MB, Osai W, Kincaid M, Wen S, Thall PF, Pettaway CA. Neoadjuvant paclitaxel, ifosfamide, and cisplatin chemotherapy for metastatic penile cancer: a phase II study. J Clin Oncol. 2010 Aug 20;28(24):3851-7. doi: 10.1200/JCO.2010.29.5477. Epub 2010 Jul 12. PMID 20625118
- [Background] Lavens N, Gupta R, Wood LA. EGFR overexpression in squamous cell carcinoma of the penis. Curr Oncol. 2010 Feb;17(1):4-6. doi: 10.3747/co.v17i1.471. No abstract available. PMID 20179797
- [Background] Andersson P, Kolaric A, Windahl T, Kirrander P, Soderkvist P, Karlsson MG. PIK3CA, HRAS and KRAS gene mutations in human penile cancer. J Urol. 2008 May;179(5):2030-4. doi: 10.1016/j.juro.2007.12.040. Epub 2008 Mar 19. PMID 18355852
- [Background] Dorff T. EGFR, TS and ERCC1 expression in penile squamous cancer. ASCO GU 2011. Not yet published.
- [Background] Valverde C.M. BRAF and KRAS mutations in penile cancer and their correlation with clinical features. ASCO GU 2011. Not yet published.
- [Background] Bonner JA, Harari PM, Giralt J, Azarnia N, Shin DM, Cohen RB, Jones CU, Sur R, Raben D, Jassem J, Ove R, Kies MS, Baselga J, Youssoufian H, Amellal N, Rowinsky EK, Ang KK. Radiotherapy plus cetuximab for squamous-cell carcinoma of the head and neck. N Engl J Med. 2006 Feb 9;354(6):567-78. doi: 10.1056/NEJMoa053422. PMID 16467544
- [Background] Cunningham D, Humblet Y, Siena S, Khayat D, Bleiberg H, Santoro A, Bets D, Mueser M, Harstrick A, Verslype C, Chau I, Van Cutsem E. Cetuximab monotherapy and cetuximab plus irinotecan in irinotecan-refractory metastatic colorectal cancer. N Engl J Med. 2004 Jul 22;351(4):337-45. doi: 10.1056/NEJMoa033025. PMID 15269313
- [Background] Pirker R, Pereira JR, Szczesna A, von Pawel J, Krzakowski M, Ramlau R, Vynnychenko I, Park K, Yu CT, Ganul V, Roh JK, Bajetta E, O'Byrne K, de Marinis F, Eberhardt W, Goddemeier T, Emig M, Gatzemeier U; FLEX Study Team. Cetuximab plus chemotherapy in patients with advanced non-small-cell lung cancer (FLEX): an open-label randomised phase III trial. Lancet. 2009 May 2;373(9674):1525-31. doi: 10.1016/S0140-6736(09)60569-9. PMID 19410716
- [Background] Baselga J, Pfister D, Cooper MR, Cohen R, Burtness B, Bos M, D'Andrea G, Seidman A, Norton L, Gunnett K, Falcey J, Anderson V, Waksal H, Mendelsohn J. Phase I studies of anti-epidermal growth factor receptor chimeric antibody C225 alone and in combination with cisplatin. J Clin Oncol. 2000 Feb;18(4):904-14. doi: 10.1200/JCO.2000.18.4.904. PMID 10673534
- [Background] Bonner JA, Harari PM, Giralt J, Cohen RB, Jones CU, Sur RK, Raben D, Baselga J, Spencer SA, Zhu J, Youssoufian H, Rowinsky EK, Ang KK. Radiotherapy plus cetuximab for locoregionally advanced head and neck cancer: 5-year survival data from a phase 3 randomised trial, and relation between cetuximab-induced rash and survival. Lancet Oncol. 2010 Jan;11(1):21-8. doi: 10.1016/S1470-2045(09)70311-0. Epub 2009 Nov 10. PMID 19897418
- [Background] Vermorken JB, Mesia R, Rivera F, Remenar E, Kawecki A, Rottey S, Erfan J, Zabolotnyy D, Kienzer HR, Cupissol D, Peyrade F, Benasso M, Vynnychenko I, De Raucourt D, Bokemeyer C, Schueler A, Amellal N, Hitt R. Platinum-based chemotherapy plus cetuximab in head and neck cancer. N Engl J Med. 2008 Sep 11;359(11):1116-27. doi: 10.1056/NEJMoa0802656. PMID 18784101
- [Background] Vermorken JB, Trigo J, Hitt R, Koralewski P, Diaz-Rubio E, Rolland F, Knecht R, Amellal N, Schueler A, Baselga J. Open-label, uncontrolled, multicenter phase II study to evaluate the efficacy and toxicity of cetuximab as a single agent in patients with recurrent and/or metastatic squamous cell carcinoma of the head and neck who failed to respond to platinum-based therapy. J Clin Oncol. 2007 Jun 1;25(16):2171-7. doi: 10.1200/JCO.2006.06.7447. PMID 17538161
- [Background] Rescigno P, Matano E, Raimondo L, Mainolfi C, Federico P, Buonerba C, Di Trolio R, D'Aniello C, Damiano V, Palmieri G, De Placido S, Di Lorenzo G. Combination of docetaxel and cetuximab for penile cancer: a case report and literature review. Anticancer Drugs. 2012 Jun;23(5):573-7. doi: 10.1097/CAD.0b013e328350ead7. PMID 22481064
- [Background] Van Cutsem E, Kohne CH, Hitre E, Zaluski J, Chang Chien CR, Makhson A, D'Haens G, Pinter T, Lim R, Bodoky G, Roh JK, Folprecht G, Ruff P, Stroh C, Tejpar S, Schlichting M, Nippgen J, Rougier P. Cetuximab and chemotherapy as initial treatment for metastatic colorectal cancer. N Engl J Med. 2009 Apr 2;360(14):1408-17. doi: 10.1056/NEJMoa0805019. PMID 19339720